CLINICAL TRIAL: NCT03266328
Title: Procedure and In-hospital Outcome of Patients Under 40 Years Old Undergoing Primary Percutaneous Coronary Intervention for Acute ST Elevated Myocardial Infarction in Assiut University
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mohamed taha galal, resident at cardiology department at assiut university hospital, Assiut University
Other Study IDs: 17100289
Record Dates: First submitted 2017-08-24; First posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1: ST elevated myocardial infarction patient presented to assiut university hospital for Primary Percutaneous Coronary Intervention (PPCI) and their age is up to 40 years old
  Interventions: Procedure: Primary Percutaneous Coronary Intervention (PPCI)
- group 2: ST elevated myocardial infarction patient presented to assiut university hospital for Primary Percutaneous Coronary Intervention (PPCI) and their age is more than 40 years old
  Interventions: Procedure: Primary Percutaneous Coronary Intervention (PPCI)

INTERVENTIONS:
Procedure: Primary Percutaneous Coronary Intervention (PPCI) — Percutaneous Coronary Intervention in patients of acute myocardial infarction diagnosed using ECG findings

SUMMARY:
Sample size of 117 patients presented with ST elevated myocardial infarction for PPCI starting from september 2017 will be divided to 2 groups, group 1 age up to 40 years old and group 2 older than 40 years then previous history and clinical data and angiographic data at PPCI and follow up in-hospital and after discharge for 3 months all these data will be compared at both groups.

DETAILED DESCRIPTION:
Myocardial infarction (MI) is a disease of middle and advanced age.

Most of the present knowledge of infarction is derived from studies in this older cohort of patients.

In fact, some clinical studies of patients with chest pain have excluded individuals under 40 years of age

Although thrombolytic therapy has been shown to improve survival in elderly AMI patients when compared with placebo, many studies have shown lower mortality rates when these patients are treated with primary percutaneous coronary intervention(PPCI) for AMI

Young adults are a relatively small portion of those having acute myocardial infarction (AMI). However they are an important group to examine with regard to risk factor modification and secondary prevention.

Previous studies have estimated that young patients of less than 40 years old make up between 2% and 6% of all AMI

young patients has different characteristics from that in the older coronary arteriography performed in young patients after myocardial infarction has identified a relatively high prevalence of angiographically normal coronary arteries.

Risk factor analysis in young AMI patients has revealed a high prevalence of current smoking, hyperlipidemia and positive family history

In addition, non-classical risk factors such as vasospastic tendencies, thrombophilic conditions and a history of Kawasaki disease have also been proposed as the causes of AMI in young patients.

PPCI is now widely accepted as a therapeutic strategy for older patients with AMI. Early, complete revascularization can salvage myocardium at risk and improve survival rates.

However on the basis of the difference in etiology of AMI, there is a possibility that the clinical effectiveness of PCI for young adults with AMI might be different from that old patients

Nevertheless, coronary artery disease has been recognized in young age groups more frequently in recent years.

It is a topic of increasing clinical interest due to the potential for premature death and long-term disability.

Aim of the study :

The purpose of the present study is to examine the clinical background, angiographic findings, acute results and in-hospital outcome of PPCI in young adults with AMI (less than 40 years) compared with those non young group (more than 40 years) .

Type of the study: case only , prospective study .Study Setting: cardiology department , assuit university hospital , assuit , Egypt

Study subjects:

1. Inclusion criteria:

   All patients with acute myocardial infarction (STEMI) : chest pain > 30 minutes and ST segment elevation in more than one lead , treated with PPCI at assuit university hospital starting from September 2017 .
2. Exclusion criteria:

   Patients undergoing elective percutaneous intervention and thrombolytic therapy.
3. Sample Size Calculation: : Sample size was calculated using Epi-info version 3 , based on previous studies , prevalence of MI in Egypt is 8.3 % , with confident level of 95 % , the sample needed for the study was estimated to be about 117

Study tools (in detail, e.g., lab methods, instruments, steps, chemicals, …):

All patient will be subjected to :

1-history taking , clinical examination & assessment of clinical risk factors of coronary heart disease as ( age , sex , family history ,DM , HTN ,smoking , addiction and type of addiction , previous ACS ,previous PCI , psychic trauma ,history of chest obstructive , renal and vascular disease , weight ,length ,BMI ,BSA , obesity , KILLIP class , ischemic time , preinfarction angina ,mode of transport 2-12 lead ECG before and after PPCI. 3-Angiongraphic findings, acute results of PPCI ( previous PCI , culprit artery , if MVD , which segment affected ,presence or absence of visible thrombus ,type of penetrating wire ,direct stenting or not ,type of the stent , name of the stent , number of stents , diameter and length of each stent , usage of thrombus aspiration , balloon dilatation ,diameter and length of the balloon ,and inflation pressure ,volume of contrast ,final TIMI flow ,presence of collaterals.

4-evaluation of PCI success (in-hospital):

a-angiographic success :( residual stenosis ≤ 30% and TIMI flow grade 3) and side branch angiographic success (residual stenosis ≤ 50% and TIMI flow grade 3)

a- procedural success : achievement of angiographic success without major clinical complication as ( death ,MI ,emergency coronary artery bypass surgery ) during hospitalization .

c- clinical success : in the short term , recovering of signs and symptoms of myocardial ischemia .

5-Therapuetic data as ( aspirin loading dose , clopidogrel loading dose ,maintenance dose and its duration , ticagrelor loading dose ,maintenance dose and its duration , usage of tirofiban intracoronary or intravenous ) 6- echocardiographic finding during admission ( EF by Simpson and M-mode , SWMA, mechanical complication ) 7-laboratory finding during admission ( total cholesterol , LDL , HDL , TG , basal creatinine , creatinine at discharge ,basal CK and CKMB , peak CK and CKMB , CK - CKMB - TNL at discharge , hemoglobin and platelet level ) 8-follow up after 3 months for ( mortality , ACS, MI , target artery revascularization ,ISR ,HF ,follow up echo EF by Simpson and M-mode , SWMA )

ELIGIBILITY:
Inclusion Criteria:

* All patients with acute myocardial infarction (STEMI): chest pain > 30 minutes and ST segment elevation in more than one lead, treated with PPCI at Assiut University Hospitals starting from September 2017.

Exclusion Criteria:

* Patients undergoing elective percutaneous intervention and thrombolytic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute myocardial infarction who receive treatment at Assiut University Hospitals in the acute setting.
Sampling Method: Probability Sample
Enrollment: 117 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
clinical outcome | 48 hours
  Evaluation of PCI success (in-hospital):
  1. angiographic success: (residual stenosis ≤ 30% and TIMI flow grade 3) and side branch angiographic success (residual stenosis ≤ 50% and TIMI flow grade 3) am
  2. procedural success: achievement of angiographic success without major clinical complication as (death, MI,emergency coronary artery bypass surgery) during hospitalization.
  3. clinical success: in the short term, recovering of signs and symptoms of myocardial ischemia.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee TH, Cook EF, Weisberg M, Sargent RK, Wilson C, Goldman L. Acute chest pain in the emergency room. Identification and examination of low-risk patients. Arch Intern Med. 1985 Jan;145(1):65-9. PMID 3970650
- [Background] Pozen MW, D'Agostino RB, Selker HP, Sytkowski PA, Hood WB Jr. A predictive instrument to improve coronary-care-unit admission practices in acute ischemic heart disease. A prospective multicenter clinical trial. N Engl J Med. 1984 May 17;310(20):1273-8. doi: 10.1056/NEJM198405173102001. PMID 6371525
- [Background] Towbin JA, Bricker JT, Garson A Jr. Electrocardiographic criteria for diagnosis of acute myocardial infarction in childhood. Am J Cardiol. 1992 Jun 15;69(19):1545-8. doi: 10.1016/0002-9149(92)90700-9. PMID 1598867
- [Background] Weinberger I, Rotenberg Z, Fuchs J, Sagy A, Friedmann J, Agmon J. Myocardial infarction in young adults under 30 years: risk factors and clinical course. Clin Cardiol. 1987 Jan;10(1):9-15. doi: 10.1002/clc.4960100104. PMID 3815921
- [Background] Chouhan L, Hajar HA, Pomposiello JC. Comparison of thrombolytic therapy for acute myocardial infarction in patients aged < 35 and > 55 years. Am J Cardiol. 1993 Jan 15;71(2):157-9. doi: 10.1016/0002-9149(93)90731-q. PMID 8421976
- [Background] Perski A, Olsson G, Landou C, de Faire U, Theorell T, Hamsten A. Minimum heart rate and coronary atherosclerosis: independent relations to global severity and rate of progression of angiographic lesions in men with myocardial infarction at a young age. Am Heart J. 1992 Mar;123(3):609-16. doi: 10.1016/0002-8703(92)90497-j. PMID 1539512
- [Background] Weaver WD, Litwin PE, Martin JS, Kudenchuk PJ, Maynard C, Eisenberg MS, Ho MT, Cobb LA, Kennedy JW, Wirkus MS. Effect of age on use of thrombolytic therapy and mortality in acute myocardial infarction. The MITI Project Group. J Am Coll Cardiol. 1991 Sep;18(3):657-62. doi: 10.1016/0735-1097(91)90784-7. PMID 1869726
- [Background] Global Use of Strategies to Open Occluded Coronary Arteries in Acute Coronary Syndromes (GUSTO IIb) Angioplasty Substudy Investigators. A clinical trial comparing primary coronary angioplasty with tissue plasminogen activator for acute myocardial infarction. N Engl J Med. 1997 Jun 5;336(23):1621-8. doi: 10.1056/NEJM199706053362301. PMID 9173270
- [Background] Zimmerman FH, Cameron A, Fisher LD, Ng G. Myocardial infarction in young adults: angiographic characterization, risk factors and prognosis (Coronary Artery Surgery Study Registry). J Am Coll Cardiol. 1995 Sep;26(3):654-61. doi: 10.1016/0735-1097(95)00254-2. PMID 7642855
- [Background] Fournier JA, Sanchez A, Quero J, Fernandez-Cortacero JA, Gonzalez-Barrero A. Myocardial infarction in men aged 40 years or less: a prospective clinical-angiographic study. Clin Cardiol. 1996 Aug;19(8):631-6. doi: 10.1002/clc.4960190809. PMID 8864336
- [Background] Imazio M, Bobbio M, Bergerone S, Barlera S, Maggioni AP. Clinical and epidemiological characteristics of juvenile myocardial infarction in Italy: the GISSI experience. G Ital Cardiol. 1998 May;28(5):505-12. PMID 9646064
- [Background] Kannel WB, Abbott RD. Incidence and prognosis of unrecognized myocardial infarction. An update on the Framingham study. N Engl J Med. 1984 Nov 1;311(18):1144-7. doi: 10.1056/NEJM198411013111802. PMID 6482932
- [Background] Warren SE, Thompson SI, Vieweg WV. Historic and angiographic features of young adults surviving myocardial infarction. Chest. 1979 Jun;75(6):667-70. doi: 10.1378/chest.75.6.667. PMID 436516
- [Background] Wolfe MW, Vacek JL. Myocardial infarction in the young. Angiographic features and risk factor analysis of patients with myocardial infarction at or before the age of 35 years. Chest. 1988 Nov;94(5):926-30. doi: 10.1378/chest.94.5.926. PMID 3180896
- [Background] Davia JE, Hallal FJ, Cheitlin MD, Gregoratos G, McCarty R, Foote W. Coronary artery disease in young patients: arteriographic and clinical review of 40 cases aged 35 and under. Am Heart J. 1974 Jun;87(6):689-96. doi: 10.1016/0002-8703(74)90412-8. No abstract available. PMID 4828802
- [Background] Thompson SI, Vieweg WV, Alpert JS, Hagan AD. Incidence and age distribution of patients with myocardial infarction and normal coronary arteriograms. Cathet Cardiovasc Diagn. 1977;3(1):1-9. doi: 10.1002/ccd.1810030102. PMID 837428
- [Background] Glover MU, Kuber MT, Warren SE, Vieweg WV. Myocardial infarction before age 36: risk factor and arteriographic analysis. Am J Cardiol. 1982 May;49(7):1600-3. doi: 10.1016/0002-9149(82)90234-x. PMID 6123253
- [Background] Waters DD, Halphen C, Theroux P, David PR, Mizgala HF. Coronary artery disease in young women: clinical and angiographic features and correlation with risk factors. Am J Cardiol. 1978 Jul;42(1):41-7. doi: 10.1016/0002-9149(78)90982-7. PMID 677035
- [Background] Salem BI, Haikal M, Zambrano A, Bollis A, Gowda S. Acute myocardial infarction with "normal" coronary arteries: clinical and angiographic profiles, with ergonovine testing. Tex Heart Inst J. 1985 Mar;12(1):1-7. PMID 15227036
- [Background] Wei JY, Bulkley BH. Myocardial infarction before age 36 years in women: predominance of apparent nonatherosclerotic events. Am Heart J. 1982 Sep;104(3):561-6. doi: 10.1016/0002-8703(82)90227-7. PMID 7113896
- [Background] Welch CC, Proudfit WL, Sheldon WC. Coronary arteriographic findings in 1,000 women under age 50. Am J Cardiol. 1975 Feb;35(2):211-5. doi: 10.1016/0002-9149(75)90003-x. PMID 1168016
- [Background] Engel HJ, Engel E, Lichtlen PR. Coronary atherosclerosis and myocardial infarction in young women--role of oral contraceptives. Eur Heart J. 1983 Jan;4(1):1-6. doi: 10.1093/oxfordjournals.eurheartj.a061365. No abstract available. PMID 6832174
- [Background] Garoufalis S, Kouvaras G, Vitsias G, Perdikouris K, Markatou P, Hatzisavas J, Kassinos N, Karidis K, Foussas S. Comparison of angiographic findings, risk factors, and long term follow-up between young and old patients with a history of myocardial infarction. Int J Cardiol. 1998 Nov 30;67(1):75-80. doi: 10.1016/s0167-5273(98)00194-6. PMID 9880203
- [Background] Williams MJ, Restieaux NJ, Low CJ. Myocardial infarction in young people with normal coronary arteries. Heart. 1998 Feb;79(2):191-4. doi: 10.1136/hrt.79.2.191. PMID 9538315
- [Background] Choudhury L, Marsh JD. Myocardial infarction in young patients. Am J Med. 1999 Sep;107(3):254-61. doi: 10.1016/s0002-9343(99)00218-1. PMID 10492319
- [Background] Doughty M, Mehta R, Bruckman D, Das S, Karavite D, Tsai T, Eagle K. Acute myocardial infarction in the young--The University of Michigan experience. Am Heart J. 2002 Jan;143(1):56-62. doi: 10.1067/mhj.2002.120300. PMID 11773912
- [Background] Suzuki A, Yamagishi M, Kimura K, Sugiyama H, Arakaki Y, Kamiya T, Miyatake K. Functional behavior and morphology of the coronary artery wall in patients with Kawasaki disease assessed by intravascular ultrasound. J Am Coll Cardiol. 1996 Feb;27(2):291-6. doi: 10.1016/0735-1097(95)00447-5. PMID 8557896
- [Background] Saigo M, Waters DD, Abe S, Biro S, Minagoe S, Maruyama I, Tei C. Soluble fibrin, C-reactive protein, fibrinogen, factor VII, antithrombin, proteins C and S, tissue factor, D-dimer, and prothrombin fragment 1 + 2 in men with acute myocardial infarction </=45 years of age. Am J Cardiol. 2004 Dec 1;94(11):1410-3. doi: 10.1016/j.amjcard.2004.07.144. PMID 15566913
- [Background] . The AMI-Kyoto Multi-Center Risk Study, a large multicenter observational study in which 15 collaborating hospitals in Kyoto Prefecture have collected demographic, procedural and outcome data on AMI patients, was established in 2000 in order to analyze this data and establish an emergency-hospital network for heart diseases in Kyoto
- [Background] Lamm G. The epidcmiology of acutc myocardial infarction in young age groups. In: Roskamm H, editor. Mw>cardial infarction at young age. Berlin:Springer-Verlag, 1981:5-12
- [Background] Burkart F, Salzmann C Angiographic findings in postinfarction patientsunder the age of 35. In ref. 2:56 60
- [Background] Motet P, Gutzwiller F, Junod B. Coronary artery disease in young adults under 35 years old: risk factors. In ref. 2:17-
- [Background] Gohlke H, Sturzenhofecker P, Thilo A, Droste C, Gornandt L, Roskamm Coronary angiographic findings and risk factors in postinfarction patients In ref. 2:61-77
- [Background] Hoit BD, Gilpin EA, Henning H, Maisel AA, Dittrich H, Carlisle J, Ross J Jr. Myocardial infarction in young patients: an analysis by age subsets. Circulation. 1986 Oct;74(4):712-21. doi: 10.1161/01.cir.74.4.712. PMID 3757185